CLINICAL TRIAL: NCT01501175
Title: Evaluation of Annual Incidence of Superficial Vein Thrombosis in the Legs
Brief Title: Incidence of Superficial Vein Thrombosis
Acronym: STEPH
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 1108036; 11.385 (Other: CCTIRS)
Record Dates: First submitted 2011-12-27; First posted 2011-12-29 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2013-02

CONDITIONS: Superficial Vein Thrombosis
Keywords: superficial vein thrombosis; Saint Etienne region
MeSH Terms: interventions — Referral and Consultation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients with suspected SVT: patients with suspected SVT and inhabitants of the Saint Etienne region
  Interventions: Other: consultation with a vascular physician

INTERVENTIONS:
Other: consultation with a vascular physician — As in usual practice, patient with suspected SVT will consult a vascular physician to diagnose SVT and eventually DVP/PE associated. Vascular physician will collect risk factors of SVT.

SUMMARY:
To date, the investigators still do not know the annual incidence of Superficial Vein Thrombosis in the legs, although the investigators do know that this pathology is frequent and the investigators can assume its incidence is greater than Deep Vein Thrombosis which is of 1 to 2 cases per year per 1,000 inhabitants. Furthermore, the high percentage of SVT with concomitant DVT and Pulmonary Embolism only concerns patients seen in vascular medicine, so it is important to re-evaluate this rate on an unselected population from general practice.

DETAILED DESCRIPTION:
The method is a prospective observational study involving all the general practitioners and vascular physicians of the Saint Etienne region, i.e. 276 general practitioners, 27 vascular physicians and 341,822 inhabitants. Any new case of symptomatic SVT in the legs suspected by the general practitioner and confirmed by compression ultrasonography by the vascular physician would be listed over one year. The confirmed SVTs, directly seen by the vascular physicians would also be listed. The incidence would be calculated by relating the total number of SVTs observed to the number of inhabitants of the Saint Etienne region. Information on whether concomitant DVT exists or not at the time of the compression ultrasonography would also be collected.

ELIGIBILITY:
Inclusion Criteria:

* inhabitants of the Saint Etienne region
* with suspected SVT
* consulting general practitioners and or vascular physicians of the Saint Etienne region

Exclusion Criteria:

* SVT not confirmed by compression ultrasonography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with suspected SVT inhabitant of the Saint Etienne region
Sampling Method: Non-Probability Sample
Enrollment: 848 (Actual)
Dates: Start 2011-11; Primary Completion 2012-11 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
symptomatic SVT | 1 year
  new case of symptomatic SVT in the legs suspected by the general practitioner and confirmed by compression ultrasonography by the vascular physician

SECONDARY OUTCOMES:
SVT risk factors | 1 year
  SVT risk factors will be collected during consultation with vascular physician. They are: varicose veins, history of thromboembolism, autoimmune disease,cancer, immobilization, recent surgery
SVT Clinical signs | 1 year
  SVT clinical signs will be collected during consultation with general practitioner and or vascular physician. They are: palpable cords, pain, erythematous area and surrounding edema.

CONTACTS AND LOCATIONS:
Overall Officials: Hervé DECOUSUS, MD PhD, Principal Investigator — CHU SAINT-ETIENNE; Paul FRAPPE, MD, Study Director — University of Saint-Etienne; Bernard TARDY, MD PhD, Study Director — CHU de Saint Etienne
Locations (7):
- France (7):
  - Cabinet D'Angiologie, Firminy
  - Ch Firminy, Firminy
  - Cabinet D'Angiologie, Saint-Chamond
  - Centre médical de Chavannes, Saint-Chamond
  - Cabinet D'Angiologie, Saint-Etienne
  - Chu Saint-Etienne, Saint-Etienne
  - Clinique Mutualiste CHirurgicale de St-Etienne, Saint-Etienne